CLINICAL TRIAL: NCT01452464
Title: A Phase IV Study to Assess the Safety of Menveo Vaccine Being Used by HMO Subjects Aged 11-21 Years of Age
Brief Title: Safety of MenACWY-CRM Vaccination in Adolescents
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V59_34OB
Record Dates: First submitted 2011-09-29; First posted 2011-10-14 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Meningococcal Disease
Keywords: observational; serogroup A, B, Y, W; meningococcal meningitis; meningococcal vaccines; safety; MenACYW-CRM; post-marketing; adolescents
MeSH Terms: conditions — Meningococcal Infections; Meningitis, Meningococcal | interventions — MenACWY-CRM vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- MenACYW-CRM vaccinated adolescents: All adolescent recipients of MenACYW-CRM vaccines during the study period. Among these, adolescents who have additionally experienced an event of interest within the 1-year observation period following vaccination will be included in the self-controlled case series.
  Interventions: Biological: MenACWY-CRM

INTERVENTIONS:
Biological: MenACWY-CRM — MenACYW-CRM vaccination received as part of routine clinical care and as registered in the vaccine records.

SUMMARY:
The purpose of this US FDA post-marketing commitment study is to evaluate the safety of MenACWY-CRM among 50.000 vaccinated adolescents within a large US Healthcare Maintenance Organization who received MenACWY-CRM vaccination as part of their routine clinical care. The pre-specified 26 events of interest are events commonly evaluated in vaccine safety studies and include certain neurological, immunological, vascular, musculoskeletal and hematologic disorders. All events are collected retrospectively.

DETAILED DESCRIPTION:
This is an observational study, vaccines administration and data that is collected is only as part of routine clinical care. Vaccinated subjects are not actively recruited.

Events of interest: Seizure, Aseptic meningitis, Bell's Palsy, Multiple Sclerosis, Guillain-Barre Syndrome, Acute disseminated encephalomyelitis, Cerebellar ataxia, Transverse myelitis, Brachial Neuritis, Hashimoto's disease, Systemic Lupus Erythematosis, Henoch Schonlein Purpura, New Onset Juvenile Diabetes Mellitus, Rheumatoid arthritis, Idiopathic Thrombocytopenic Purpura, Iridocyclitis, Acute glomerulonephritis, Nephrotic syndrome, Grave's disease, Autoimmune hemolytic anemia, Myasthenia Gravis, New onset asthma, Allergic urticaria, Anaphylaxis, Meningococcal Disease, Suicide attempt.

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in the HMO for at least 6 months prior to vaccination
2. Between the ages of 11 and 21 years (inclusive - i.e. has not reached their 22nd birthday) at the time of the vaccination.
3. Received the vaccine during the study period

Exclusion Criteria:

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population is selected from the Health Maintenance Organization population of the Kaiser Permanente Southern California (KPSC) HMO in Pasadena, CA, USA.
Sampling Method: Non-Probability Sample
Enrollment: 55397 (Actual)
Dates: Start 2011-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Relative incidence (RI) for an Event of Interest (EOI) is calculated using the self controlled case series method. RI is the ratio of the incidence of an EOI in a pre-specified, event-specific risk window relative to the incidence in the control period. | Observational period of 1 year following date of vaccination of that individual.

SECONDARY OUTCOMES:
Frequency (n,%) of each EOI is calculated. | Observational period of 1 year following date of vaccination of that individual.
Incidence (n/person yrs) of each EOI is calculated. | Observational period of 1 year following date of vaccination of that individual.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (3):
- United States (3):
  - Riverside Medical Center Campus, 10800 Magnolia Ave, Riverside, California
  - San Diego Medical Center Campus, 4647 Zion Ave 92120, San Diego, California
  - Fontana Medical Center Campus, Valley Annex, 16994 E. Valley Blvd., Fontana, California